CLINICAL TRIAL: NCT03497182
Title: Study to Assess Feasibility of Sepsis, Severe Sepsis and Septic Shock Detection by Breath Analysis
Brief Title: Sepsis, Severe Sepsis and Septic Shock Detection by Breath Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landon Pediatric Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Study 177: ZNose
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Breath sample collection (Experimental)
  Interventions: Device: Breath sample collection

INTERVENTIONS:
Device: Breath sample collection — Subject exhales into breath collection container.

SUMMARY:
Breath samples will be collected from patients suspected of sepsis/severe sepsis or septic shock according to hospital sepsis screening criteria in the Emergency Department.

DETAILED DESCRIPTION:
Breath samples will be collected from patients suspected of sepsis that meet the criteria in the hospital's Sepsis Patient Management Protocol for blood lactate point of care testing. The breath samples will be collected from the patient by the Respiratory Therapist (RT) at the time of blood sample collection for the blood lactate test.

The breath samples will be analyzed via gas chromatography-surface acoustic wave spectroscopy for detection of a pattern of volatile organic compounds (VOCs). Multivariate analysis will be performed on breath sample data to determine feasibility of associating a unique VOC pattern with septic/severe septic/septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* admitted to Emergency Department
* suspected of sepsis according to hospital screening criteria; point of care blood lactate test performed
* age 18 or older

Exclusion Criteria:

* member of Vulnerable Patient Population
* unable to complete Patient Informed Consent process/document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-10-06 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Volatile Organic Compound (VOC) Pattern | five minutes
  Detection of a unique pattern of Volatile Organic Compounds (VOCs) in the breath samples of patients confirmed as having sepsis/severe sepsis/septic shock differentiated from subjects confirmed as not septic.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Landon, Principal Investigator — Director Pediatrics
Locations (1):
- Ventura County Medical Center, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No